CLINICAL TRIAL: NCT00235378
Title: Gene Mapping in Women With SLE
Brief Title: Genetic Study of Lupus Patients and Their Families
Status: Completed | Type: Observational
Sponsor: Oklahoma Medical Research Foundation (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01AR043274 (NIH); R01AR043274 (NIH)
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: SLE patients
- 2: Unaffected family members of SLE patients
- 3: Control participants

SUMMARY:
The purpose of this study is to perform genetic testing in and to collect information from families affected by lupus in order to identify the genetic factors associated with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
Little is known about the genetic factors that predispose people to developing SLE. Genes in patients with SLE may provide clues about SLE's pathogenesis. This study will compare genes from SLE patients, their unaffected family members, and control participants. Travel to the study site is not required.

In this study, blood samples will be collected from people diagnosed with SLE, their unaffected family members, and condition-matched controls. Participants will be asked questions about their health and will provide a small blood sample. Participants will also be asked to provide written permission for release of medical information, so that their disease status can be verified through medical record review or through consultation with their doctors. Study personnel may contact participants in the future for follow-up questions and additional blood draws, if the participant agrees.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE OR a family member of participant diagnosed with SLE

Exclusion Criteria:

* Pregnancy or breastfeeding

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants include SLE patients, their unaffected family members, and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 2356 (Actual)
Dates: Start 1996-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W. Behrens, MD, Principal Investigator — University of Minnesota; Patrick Gaffney, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Baechler EC, Batliwalla FM, Karypis G, Gaffney PM, Ortmann WA, Espe KJ, Shark KB, Grande WJ, Hughes KM, Kapur V, Gregersen PK, Behrens TW. Interferon-inducible gene expression signature in peripheral blood cells of patients with severe lupus. Proc Natl Acad Sci U S A. 2003 Mar 4;100(5):2610-5. doi: 10.1073/pnas.0337679100. Epub 2003 Feb 25. PMID 12604793
- [Background] Gillett CD, Langefeld CD, Williams AH, Ortmann WA, Graham RR, Rodine PR, Selby SA, Gaffney PM, Behrens TW, Moser KL. Fine mapping chromosome 16q12 in a collection of 231 systemic lupus erythematosus sibpair and multiplex families. Genes Immun. 2005 Feb;6(1):19-23. doi: 10.1038/sj.gene.6364145. PMID 15538391
- [Background] Graham RR, Ortmann WA, Langefeld CD, Jawaheer D, Selby SA, Rodine PR, Baechler EC, Rohlf KE, Shark KB, Espe KJ, Green LE, Nair RP, Stuart PE, Elder JT, King RA, Moser KL, Gaffney PM, Bugawan TL, Erlich HA, Rich SS, Gregersen PK, Behrens TW. Visualizing human leukocyte antigen class II risk haplotypes in human systemic lupus erythematosus. Am J Hum Genet. 2002 Sep;71(3):543-53. doi: 10.1086/342290. Epub 2002 Jul 26. PMID 12145745
- [Background] Kyogoku C, Langefeld CD, Ortmann WA, Lee A, Selby S, Carlton VE, Chang M, Ramos P, Baechler EC, Batliwalla FM, Novitzke J, Williams AH, Gillett C, Rodine P, Graham RR, Ardlie KG, Gaffney PM, Moser KL, Petri M, Begovich AB, Gregersen PK, Behrens TW. Genetic association of the R620W polymorphism of protein tyrosine phosphatase PTPN22 with human SLE. Am J Hum Genet. 2004 Sep;75(3):504-7. doi: 10.1086/423790. Epub 2004 Jul 23. PMID 15273934
- [Background] Wakeland EK, Liu K, Graham RR, Behrens TW. Delineating the genetic basis of systemic lupus erythematosus. Immunity. 2001 Sep;15(3):397-408. doi: 10.1016/s1074-7613(01)00201-1. PMID 11567630